CLINICAL TRIAL: NCT01531972
Title: A Phase 1, Open-Label, Single-photon Emission Computed Tomography (SPECT) Study to Evaluate Serotonin and Dopamine Transporter Occupancy After Multiple Dose Administration of SEP-228432 to Achieve Steady State in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SEP432-102
Record Dates: First submitted 2012-02-08; First posted 2012-02-13 (Estimated); Last update posted 2013-12-09 (Estimated); Status verified 2013-12

CONDITIONS: Healthy
Keywords: Single-photon Emission Computed Tomography; Healthy Volunteers; Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- SEP-228432 (Cohort 1) (Experimental): Subjects will receive 40 mg of SEP-228432 (titration) orally once per day for 3 days; followed by (steady state) at a dose of 200 mg orally once per day for 5 days.
  Interventions: Drug: SEP-228432
- SEP-228432 (Cohort 2) (Experimental): Subjects will receive 40 mg of SEP-228432 (titration) orally once per day for 3 days followed by a dose (TBD) of SEP 228432 ≤ 300mg, orally once per day for 5 days.
  Interventions: Drug: SEP-228432
- SEP-228432 (Cohort 3) (Experimental): Subjects will receive 40 mg of SEP-228432 (titration) 40 mg of SEP 228432 orally once per day for 3 days followed by a dose (TBD) of SEP 228432 ≤ 300mg, orally once per day for 5 days.
  Interventions: Drug: SEP-228432

INTERVENTIONS:
Drug: SEP-228432 — 40 mg, orally, once daily for 3 days followed by 200 mg orally, once daily for 5 days
  Arms: SEP-228432 (Cohort 1)
Drug: SEP-228432 — 40 mg orally once daily for 3 days followed by ≤ 300mg, orally once daily for 5 days
  Arms: SEP-228432 (Cohort 2); SEP-228432 (Cohort 3)

SUMMARY:
This is an open-label study investigating the relationship between SEP-228432 and SEP-228431 (the active metabolite of SEP-228432) plasma concentrations, SERT occupancy, and DAT occupancy, both measured by SPECT imaging.

DETAILED DESCRIPTION:
This is an open-label study investigating the relationship between SEP-228432 and SEP-228431 (the active metabolite of SEP-228432) plasma concentrations, SERT occupancy, and DAT occupancy, both measured by SPECT imaging using [123I]-2β-carbomethoxy-3β-(4-iodophenyl) tropane ([123I] β -CIT). Up to 3 sequential cohorts of 8 subjects each will have multiple dose administrations of SEP-228432. The target dose for the first cohort will be 200 mg. Dose selection for the remaining cohorts will be based on preliminary review of all available relevant data from prior dosing cohort(s).

ELIGIBILITY:
Inclusion Criteria:

* Subject must give written informed consent prior to participation in the study.
* Subject must be willing and able to comply with the study procedures and visit schedules and must be able to follow verbal and written instructions.
* Male and female subjects between 18-50 years of age (inclusive) at the time of signing consent.
* Subject must be judged to be in a condition of general good health (defined as the absence of any clinically relevant abnormalities as determined by the investigator), based on screening medical and psychiatric histories, physical examination, neurological examination, vital signs, clinical laboratory values (hematology, chemistry, and urinalysis), and a 12-lead ECG.
* Subject, if female, must have a negative serum pregnancy test at screening. All subjects must be instructed to and agree to avoid pregnancy during the study and must be using an acceptable method of birth control: An oral contraceptive, an intrauterine device (IUD), implantable contraceptive, transdermal or injectable contraceptive for at least 30 days prior to screening and will continue its use throughout the study and for 30 days following study participation. Barrier method of contraception, eg, condom and/or diaphragm with spermicide while participating in the study. Abstinence.
* Subject must be willing to stay within the residential facility for the required period and must be willing to attend up to 3 additional outpatient visits.
* Subject's body mass index (BMI) must be at least 16 kg/m2 but no more than 32 kg/m2.
* Subject must be willing to refrain from strenuous activity during the course of the study.

Exclusion Criteria:

* Subject has poor venous access that would cause difficulty for collecting blood samples.
* Subject with a history of exposure to any radiation ≥ 15 mSv/year (eg, occupational or radiation therapy) within the previous year.
* Subject has participated in an investigational drug study and received investigational drug within 30 days prior to signing informed consent (with the exception of previous SPECT imaging studies where the only investigational drug administered was a radiotracer), or is currently participating in another clinical trial.
* Subject has any clinically significant unstable medical condition or any clinically significant chronic disease. Subject with evidence or history of a clinically significant hematological (including deep vein thrombosis) or bleeding disorder, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (except for untreated, asymptomatic allergies at time of dosing).
* Subject has a history of severe or multiple allergic reactions to medications.
* Subject has a history of hospitalization within 45 days prior to signing informed consent.
* Subject has a positive test for Hepatitis B surface antigen, Hepatitis C antibody, human immunodeficiency virus (HIV)-1, or HIV-2 antibody, or has a history of a positive result.
* Subject has a presence or history of a medically diagnosed, clinically significant psychiatric disorder (including mental retardation).
* Female subject who is pregnant or lactating.
* Subject has a history of cancer (exception: basal cell carcinoma in remission).
* Subject has experienced significant blood loss (≥ 473 mL) or donated blood within 60 days prior to signing informed consent; has donated plasma within 72 hours prior to signing informed consent; or intends to donate plasma or blood or undergo elective surgery during study participation or within 60 days after the last study visit.
* Subject has a history of substance abuse or drug abuse within 12 months prior to signing informed consent or a positive drug screen at Visit 1.
* Subject has a history of tobacco dependency or has used tobacco or nicotine within 30 days prior to signing informed consent (including pipe, cigar, patch, chewing tobacco, spray, inhaler, or gum) or a positive urine cotinine test at Visit 1.
* Subject has a history of regular alcohol consumption exceeding 7 drinks/week for women or 14 drinks/week for men (1 drink = 5 ounces of wine or 12 ounces of beer or 1.5 ounces of hard liquor) within 6 months prior to signing informed consent.
* Subject consumes more than 180 mg of caffeine per day (3 cups of coffee or equivalent in caffeinated beverages).
* Subject has a disorder or history of a condition that may interfere with drug absorption, distribution, metabolism, or excretion or a clinically significant abnormality of the hepatic or renal system, or a history of malabsorption, or previous gastrointestinal surgery (eg, cholecystectomy, vagotomy, bowel resection, or any surgical procedure) that could affect drug absorption or metabolism, gastrointestinal motility, or pH.
* Subject has a clinically significant abnormal 12-lead ECG that may jeopardize the subject's ability to complete the study or a Screening 12-lead ECG demonstrating any one of the following: heart rate > 100 beats per minute (bpm), QRS > 120 ms, QTc > 450 ms, or PR > 220 ms as determined by the investigator using the core laboratory ECG interpretation report.
* Subject has used prescription or non-prescription drugs, vitamins, dietary or herbal supplements within 14 days prior to signing informed consent. Enzyme-inducing herbal supplements (eg, Metabolife™) must have been discontinued at least 30 days prior to signing informed consent.
* Subject previously received study drug in this study.
* Subject is a staff member or the relative of a staff member.
* Subject is in the opinion of the investigator, unsuitable in any other way to participate in this study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2012-02; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
SERT and DAT occupancy (% occupancy) achieved at steady-state concentrations of SEP-228432 and SEP-228431 in healthy subjects. | Day 8 and 9
  SERT and DAT occupancy (% occupancy) achieved at steady-state concentrations of SEP-228432 and SEP-228431 in healthy subjects.

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs). | Up to Day 16
  Incidence of treatment-emergent adverse events (TEAEs).

CONTACTS AND LOCATIONS:
Locations (1):
- Molecular NeuroImaging, New Haven, Connecticut, United States